CLINICAL TRIAL: NCT00536133
Title: Role of Zinc in Recurrent Acute Lower Respiratory Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jawaharlal Nehru Medical College (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Dr Ubaid Hameed Shah, Jawaharlal Nehru medical college, A.M.U, Aligarh, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MDPG05/01
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Acute Respiratory Infections
Keywords: zinc; aute lower respiratory infections
MeSH Terms: interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc group (Experimental): children with recurrent acute lower respiratory infections receiving zinc supplementation
  Interventions: Drug: Zinc
- Placebo group (Placebo Comparator): children with recurrent acute lower respiratory infections receiving placebo syrup
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Zinc — 5 ml of syrup containing zinc gluconate equivalent to 10 mg of elemental zinc per day for 60 days
  Arms: Zinc group
Other: placebo — 5 ml of syrup, identical in taste, color and consistency to the syrup given to zinc group, but containing no zinc
  Arms: Placebo group

SUMMARY:
Acute respiratory infections (ARIs) are the most frequent illnesses globally. Despite advances in the recognition and management ARIs, these account for over 20% of all child deaths globally.Trace mineral deficiencies have long been implicated in causation and consequences of many diseases. The importance of adequate zinc intake in human health is well documented and zinc deficiency is a large public health problem, especially among children in developing countries.Various studies suggest that zinc-deficient populations are at increased risk of developing diarrhoeal diseases, respiratory tract infections and growth retardation.Among the individual interventions zinc supplementation with universal coverage ranks 5th in preventing under five mortality in India, preceded only in order by breast feeding; complementary feeding; clean delivery; Hib vaccination; and clean water, sanitation and hygiene.Numerous studies have examined the association between child mortality and zinc deficiency. A number of randomized controlled trials evaluating effect of zinc supplementation have found the intervention to be beneficial in reducing ARI and diarrhoeal mortality and morbidity but few studies have found beneficial effect in diarrhea and no or even contrasting effects on morbidity pattern of acute respiratory infections. Whereas role of zinc in diarrhea is now a well established and specific guidelines and recommendations have been given for zinc supplementation in diarrhea, role of zinc in acute respiratory infections is controversial. The contrasting effect of zinc on diarrhoea and acute lower respiratory infection as reported in several studies is a public health concern, because zinc supplementation is carried out in many nutrition rehabilitation units. Further in many of randomized control trials supplement syrups also contained other vitamins, including vitamin A, known to have effect on respiratory morbidity. Most of the trials evaluating effect of zinc on respiratory morbidity and mortality are community based and children with well known causes of recurrent acute lower respiratory infections have not been excluded from the study pool.

Hence the current study was planned to bridge this gap of information and attempts to detect the role of zinc using "zinc only preparations" in reducing respiratory morbidity in children aged 6 to 59 months with recurrent acute lower respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 59 months with documented recurrent acute lower respiratory infection i.e., more than two episodes of ALRI in one year or more than three episodes in any time frame.

Exclusion Criteria:

* Children with congenital heart diseases
* Children with congenital anomalies which can cause recurrent chest infection
* Children with Tuberculosis
* Children with bronchial asthma or hyperactive airway disease
* Children with WZS < -2 of HZS < -2 as per WHO standards
* Children with any diarrhoeal episode in past 3 months
* Children having receive any zinc supplementation in past 3 months
* Children who did not turn up on follow up and could not be contacted were excluded from the study.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
change in mean serum zinc level; Number of episodes of ALRI per child ALRI free days per child per year; | six months

SECONDARY OUTCOMES:
Diarrhoeal episodes per child; morbidity free days per child; mean hospitalization days; change in Weight for age and height for age z scores | six months

CONTACTS AND LOCATIONS:
Overall Officials: Mohd A Malik, MD, Study Director — Professor, Department of pediatrics, Jawaharlal nehru Medical College, A.M.U, Aligarh; Ubaid H Shah, MD, Principal Investigator — Jawaharlal Nehru Medical College
Locations (1):
- Jawaharlal Nehru Medical College, Aligarh Muslim University, Aligarh, Uttar Pradesh, India

REFERENCES:
- [Background] Black RE, Morris SS, Bryce J. Where and why are 10 million children dying every year? Lancet. 2003 Jun 28;361(9376):2226-34. doi: 10.1016/S0140-6736(03)13779-8. PMID 12842379
- [Background] Caufield L, Black R. Zinc deficiency. In: Ezzati M, Lopez AD, Rodgers A, Murray C, eds. Comparative Quantification of Health Risks: Global and Regional Burden of Disease Attributable to Selected Major Risk Factors. Geneva, Switzerland: World Health Organization; 2004:257-259
- [Background] Bhatnagar S, Natchu UC. Zinc in child health and disease. Indian J Pediatr. 2004 Nov;71(11):991-5. doi: 10.1007/BF02828114. PMID 15572819
- [Background] Ruel MT, Rivera JA, Santizo MC, Lonnerdal B, Brown KH. Impact of zinc supplementation on morbidity from diarrhea and respiratory infections among rural Guatemalan children. Pediatrics. 1997 Jun;99(6):808-13. doi: 10.1542/peds.99.6.808. PMID 9164774
- [Background] Rahman MM, Vermund SH, Wahed MA, Fuchs GJ, Baqui AH, Alvarez JO. Simultaneous zinc and vitamin A supplementation in Bangladeshi children: randomised double blind controlled trial. BMJ. 2001 Aug 11;323(7308):314-8. doi: 10.1136/bmj.323.7308.314. PMID 11498488
- [Background] Sazawal S, Black RE, Jalla S, Mazumdar S, Sinha A, Bhan MK. Zinc supplementation reduces the incidence of acute lower respiratory infections in infants and preschool children: a double-blind, controlled trial. Pediatrics. 1998 Jul;102(1 Pt 1):1-5. doi: 10.1542/peds.102.1.1. PMID 9651405
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Effect of routine zinc supplementation on pneumonia in children aged 6 months to 3 years: randomised controlled trial in an urban slum. BMJ. 2002 Jun 8;324(7350):1358. doi: 10.1136/bmj.324.7350.1358. PMID 12052800
- [Derived] Shah UH, Abu-Shaheen AK, Malik MA, Alam S, Riaz M, Al-Tannir MA. The efficacy of zinc supplementation in young children with acute lower respiratory infections: a randomized double-blind controlled trial. Clin Nutr. 2013 Apr;32(2):193-9. doi: 10.1016/j.clnu.2012.08.018. Epub 2012 Aug 31. PMID 22981241